CLINICAL TRIAL: NCT03143218
Title: A Phase IIIB Comparative Trial of Seasonal Vaccination With the Malaria Vaccine RTS,S/AS01, Seasonal Malaria Chemoprevention and of the Two Interventions Combined
Brief Title: Seasonal Malaria Vaccination (RTS,S/AS01) and Seasonal Malaria Chemoprevention (SP/AQ)
Acronym: RTSS-SMC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ITDCZJ29 - Greenwood
Record Dates: First submitted 2017-03-22; First posted 2017-05-08 (Actual); Results first posted 2022-01-28 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Malaria,Falciparum; Children, Only
Keywords: Malaria; Seasonal vaccination; Seasonal chemoprevention
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — RTS,S-AS01 vaccine; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Intervention Model Description: A double-blind, individually randomised trial to compare the incidence of clinical episodes of malaria across three study arms:
  1. Seasonal vaccination with the malaria vaccine RTS,S/AS01
  2. Seasonal malaria chemoprevention with SP/AQ
  3. Combination of these two interventions
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMC with SP+AQ (Active Comparator): Administration of RABIPUR® in Year 1 and Hepatitis A vaccine in Year 2 and 3, followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1,2 and 3.
  Interventions: Biological: RABIPUR®; Drug: SMC with SP+AQ
- RTS,S/AS01 (Active Comparator): Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with placebo in Year 1,2 and 3.
  Interventions: Biological: RTS,S/AS01; Drug: SMC placebo
- RTS,S/AS01 PLUS SMC with SP+AQ (Active Comparator): Administration of the malaria vaccine RTS,S/AS01 followed by 4 cycles of SMC with sulphadoxine/pyrimethamine plus amodiaquine in Year 1,2 and 3.
  Interventions: Biological: RTS,S/AS01; Drug: SMC with SP+AQ

INTERVENTIONS:
Biological: RABIPUR® — Year 1 (2017) Three doses of rabies vaccine (April, May, June) Year 2 and 3 (2018/19) One dose of Hepatitis A vaccine (June)
  Arms: SMC with SP+AQ
Biological: RTS,S/AS01 — Year 1 (2017) Three doses of RTSS/AS01 (April, May, June) Year 2 and 3 (2018/19) One booster dose of RTSS/AS01 (June)
  Arms: RTS,S/AS01; RTS,S/AS01 PLUS SMC with SP+AQ
Drug: SMC with SP+AQ — Year 1, 2 and 3(2017/18/19) Four cycles of SMC (SP+AQ) during the malaria transmission season One cycle of SMC for children above one year of age consisting of sulphadoxine - pyrimethamin (SP) 500mg/25 mg, and amodiaquine (AQ) 150mg on day 1, and AQ 150mg on days 2 and 3. Infants will receive half of these doses.
  Arms: RTS,S/AS01 PLUS SMC with SP+AQ; SMC with SP+AQ
Drug: SMC placebo — Year 1, 2 and 3(2017/18/19) Four cycles of SMC placebo during the malaria transmission season
  Arms: RTS,S/AS01

SUMMARY:
A double-blind, individual randomised trial will be undertaken in 6000 children under the age of five years living in areas of Burkina Faso or Mali where the transmission of malaria is intense and highly seasonal to determine whether the malaria vaccine RTS,S/AS01 is (a) as effective as SMC with SP + AQ in preventing clinical malaria (b) provides additional, useful protection when given together with SMC. The primary trial end-point will be the incidence of clinical episodes of malaria detected by passive case detection.

DETAILED DESCRIPTION:
The RTS,S/AS01 malaria vaccine is a recombinant protein vaccine in which the fusion protein RTS (containing parts of the circumsporozoite protein (CSP) of Plasmodium falciparum fused to hepatitis B surface antigen (HBsAg)) is co-expressed in yeast together with free HBsAg (S) to form a virus like particle (RTS,S); it is given with the powerful adjuvant AS01. RTS,S/AS01 induces a strong antibody response to the P. falciparum CSP and high titres of anti-CSP antibody are associated with protection. Following a long process of development, a phase 3 study of RTS,S/AS01 conducted in 15,439 children in 7 countries in Africa showed that three doses of RTS,S/AS01 given with a one month interval between doses, followed by a fourth dose 18 months post dose 3, gave 36.5 % [95% CI 31,41%] protection against clinical attacks of malaria when given to young children aged 5-17 months who were followed for 48 months; efficacy was less when given to infants at the age of 6-12 weeks. RTS,S/AS01 provides a high level of protection during the first three months after vaccination, modelled to be about 70% in the phase 3 trial, a level of initial efficacy similar to that observed in an earlier phase 2 trial in Gambian adults. However, efficacy wanes progressively over the following months. A subsequent dose given 18 months after the primary series restores some but not all of the efficacy seen immediately after the primary series. In July 2015, the European Medicines Agency reviewed efficacy and safety data on RTS.S/AS01 and concluded that the risk benefit balance favoured the vaccine and gave a positive opinion on its use in children aged 6 weeks to 17 months. The World Health Organization (WHO) Strategic Advisory Group of Experts (SAGE) committee reviewed the vaccine's efficacy and safety in October 2015 and made a number of recommendations on its further evaluation. These included the pilot implementation of RTS,S/AS01 in children aged 5-17 months in 3-5 settings with moderate-to-high malaria transmission intensity, with a preference for areas where SMC is not being delivered, and evaluation of alternative approaches to deployment of the vaccine. Recent evidence from challenge studies conducted in American adult volunteers suggests that a higher level of protection can be obtained when the third dose of the priming schedule is reduced to one fifth of the usual amount and delayed until approximately 6 months post dose 2, and when a reduced dose is used for boosting. In these studies, a vaccine efficacy of 86% was achieved three weeks following priming and 90% efficacy following boosting with a fractional dose. This encouraging result is now being followed in further studies.

SMC involves monthly administration of an antimalarial drug or drug combination in a full therapeutic course to children on three of four occasions during the period of highest risk of malaria infection. Studies undertaken in several countries in West Africa, including Burkina Faso and Mali, have shown that SMC with sulphadoxine/pyrimethamine (SP) and amodiaquine (AQ) is highly effective in areas where the transmission of malaria is markedly seasonal, reducing the incidence of severe and uncomplicated malaria by up to 80%. SMC with a combination of SP and AQ is safe, with no serious drug related adverse event being reported after administration of over 800,000 courses in Senegal. Recent studies have defined the areas where SMC would be an appropriate intervention based on the seasonality and incidence of malaria. These include most of the Sahel and sub-Sahel, population approximately 200 million, and possibly other areas in southern and eastern Africa. A Technical Expert Group of the WHO reviewed all the available evidence on the efficacy and safety of SMC in May 2011 and recommended SMC with SP+AQ in areas of the Sahel and sub-Sahel with highly seasonal transmission. This recommendation was endorsed by the WHO Malaria Policy Advisory Committee (MPAC) in February 2012. Most countries in the Sahel and sub-Sahel region have incorporated SMC, along with other malaria control interventions in their strategic malaria control plan and the implementation of SMC at scale is in progress in many countries in this region through the UNITAID supported SMC ACCESS programme and the support of other major donor organisations. Preliminary evaluation suggests that SMC is providing about 50% protection against clinical malaria when delivered through a national programme (http://www.malariaconsortium.org/pages/access-smc.htm).

SMC is effective but its delivery is demanding on the recipient and provider, requiring four contacts each malaria transmission season if anti-malarials are given to mothers to administer at home and 12 contacts if directly observed treatment is employed. In addition, SMC is threatened by the emergence of resistance to SP and AQ and there are currently no other combinations of licensed antimalarials that could be used to replace them. It is likely to be 5-10 years before novel antimalarials under development could be deployed for SMC. In contrast to SMC, seasonal vaccination with RTS,S/AS01 would require only one visit each transmission season after priming. RTS,S/AS01 may be a little less effective than SMC during the malaria transmission season but this may be balanced by provision of protection during the dry season, when some malaria transmission still occurs and when SMC would provide no benefit. There is, therefore, a need for a comparative study of these two interventions. In some areas where SMC is currently being deployed, and other malaria control interventions such as long-lasting insecticide treated nets used widely, the incidence of malaria in young children remains high (0.4 episodes per year in children under the age of five years in SMC recipients in Burkina Faso). Thus, determining whether RTS,S/AS01 would provide added, useful protection to SMC in such situations is also important. It might also be able to protect some children who, because of side effects, are unable or unwilling to take SMC.

Although the European Medicines Agency has given a positive opinion on RTS,S/AS01, it is not yet certain how this partially effective malaria vaccine can be used most effectively. Three, large-scale pilot implementation studies are being planned by WHO but it is unlikely that, following WHO recommendations, any of these will be conducted in a country where SMC is being delivered. The WHO recommendations on RTS,S/AS01 indicate the need for research on alternative approaches to the delivery of this vaccine. Exploration of the potential of the vaccine to prevent seasonal malaria, taking advantage of its high but rapidly waning efficacy, meets this recommendation and is, therefore, timely.

ELIGIBILITY:
Inclusion Criteria:

* The child is a permanent resident of the study area and likely to remain a resident for the duration of the trial
* The child is 5 - 17 months of age at the time of first vaccination
* A parent or legally recognised guardian provides informed consent for the child to join the trial

Exclusion Criteria:

* The child is a transient resident in the study area
* The child is in care
* The age of the child is outside the stipulated range
* The child has a history of an adverse reaction to SP or AQ
* The child has a serious underlying illness, including known HIV infection, unless this is well controlled by treatment, or severe malnutrition (weight for age or mid arm circumference Z scores < 3 SD)
* The child is known to have an immune deficiency disease or is receiving an immunosuppressive drug
* The child has previously received a malaria vaccine.
* The child is enrolled in another malaria intervention trial
* The parents or guardians do not provide informed consent

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5920 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, Professor, Study Director — Malaria Research & Training Center, Bamako; Jean Bosco Ouedraogo, Professor, Study Director — Institut de Recherche en Sciences de la Santé, Direction Régionale de l'Ouest (IRSS-DRO)
Locations (2):
- Institut de Recherche en Sciences de la Santé, Direction Régionale de l'Ouest, Ouagadougou, Burkina Faso
- Malaria Research & Training Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the LSHTM Data Compass system

REFERENCES:
- [Background] Cohen J, Nussenzweig V, Nussenzweig R, Vekemans J, Leach A. From the circumsporozoite protein to the RTS, S/AS candidate vaccine. Hum Vaccin. 2010 Jan;6(1):90-6. doi: 10.4161/hv.6.1.9677. Epub 2010 Jan 30. PMID 19806009
- [Background] White MT, Verity R, Griffin JT, Asante KP, Owusu-Agyei S, Greenwood B, Drakeley C, Gesase S, Lusingu J, Ansong D, Adjei S, Agbenyega T, Ogutu B, Otieno L, Otieno W, Agnandji ST, Lell B, Kremsner P, Hoffman I, Martinson F, Kamthunzu P, Tinto H, Valea I, Sorgho H, Oneko M, Otieno K, Hamel MJ, Salim N, Mtoro A, Abdulla S, Aide P, Sacarlal J, Aponte JJ, Njuguna P, Marsh K, Bejon P, Riley EM, Ghani AC. Immunogenicity of the RTS,S/AS01 malaria vaccine and implications for duration of vaccine efficacy: secondary analysis of data from a phase 3 randomised controlled trial. Lancet Infect Dis. 2015 Dec;15(12):1450-8. doi: 10.1016/S1473-3099(15)00239-X. Epub 2015 Sep 2. PMID 26342424
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of RTS,S/AS01 malaria vaccine with or without a booster dose in infants and children in Africa: final results of a phase 3, individually randomised, controlled trial. Lancet. 2015 Jul 4;386(9988):31-45. doi: 10.1016/S0140-6736(15)60721-8. Epub 2015 Apr 23. PMID 25913272
- [Background] Bojang KA, Milligan PJ, Pinder M, Vigneron L, Alloueche A, Kester KE, Ballou WR, Conway DJ, Reece WH, Gothard P, Yamuah L, Delchambre M, Voss G, Greenwood BM, Hill A, McAdam KP, Tornieporth N, Cohen JD, Doherty T; RTS, S Malaria Vaccine Trial Team. Efficacy of RTS,S/AS02 malaria vaccine against Plasmodium falciparum infection in semi-immune adult men in The Gambia: a randomised trial. Lancet. 2001 Dec 8;358(9297):1927-34. doi: 10.1016/S0140-6736(01)06957-4. PMID 11747915
- [Background] Regules JA, Cicatelli SB, Bennett JW, Paolino KM, Twomey PS, Moon JE, Kathcart AK, Hauns KD, Komisar JL, Qabar AN, Davidson SA, Dutta S, Griffith ME, Magee CD, Wojnarski M, Livezey JR, Kress AT, Waterman PE, Jongert E, Wille-Reece U, Volkmuth W, Emerling D, Robinson WH, Lievens M, Morelle D, Lee CK, Yassin-Rajkumar B, Weltzin R, Cohen J, Paris RM, Waters NC, Birkett AJ, Kaslow DC, Ballou WR, Ockenhouse CF, Vekemans J. Fractional Third and Fourth Dose of RTS,S/AS01 Malaria Candidate Vaccine: A Phase 2a Controlled Human Malaria Parasite Infection and Immunogenicity Study. J Infect Dis. 2016 Sep 1;214(5):762-71. doi: 10.1093/infdis/jiw237. Epub 2016 Jun 13. PMID 27296848
- [Background] Wilson AL; IPTc Taskforce. A systematic review and meta-analysis of the efficacy and safety of intermittent preventive treatment of malaria in children (IPTc). PLoS One. 2011 Feb 14;6(2):e16976. doi: 10.1371/journal.pone.0016976. PMID 21340029
- [Background] Dicko A, Diallo AI, Tembine I, Dicko Y, Dara N, Sidibe Y, Santara G, Diawara H, Conare T, Djimde A, Chandramohan D, Cousens S, Milligan PJ, Diallo DA, Doumbo OK, Greenwood B. Intermittent preventive treatment of malaria provides substantial protection against malaria in children already protected by an insecticide-treated bednet in Mali: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000407. doi: 10.1371/journal.pmed.1000407. PMID 21304923
- [Background] Konate AT, Yaro JB, Ouedraogo AZ, Diarra A, Gansane A, Soulama I, Kangoye DT, Kabore Y, Ouedraogo E, Ouedraogo A, Tiono AB, Ouedraogo IN, Chandramohan D, Cousens S, Milligan PJ, Sirima SB, Greenwood B, Diallo DA. Intermittent preventive treatment of malaria provides substantial protection against malaria in children already protected by an insecticide-treated bednet in Burkina Faso: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000408. doi: 10.1371/journal.pmed.1000408. PMID 21304925
- [Background] NDiaye JL, Cisse B, Ba EH, Gomis JF, Ndour CT, Molez JF, Fall FB, Sokhna C, Faye B, Kouevijdin E, Niane FK, Cairns M, Trape JF, Rogier C, Gaye O, Greenwood BM, Milligan PJ. Safety of Seasonal Malaria Chemoprevention (SMC) with Sulfadoxine-Pyrimethamine plus Amodiaquine when Delivered to Children under 10 Years of Age by District Health Services in Senegal: Results from a Stepped-Wedge Cluster Randomized Trial. PLoS One. 2016 Oct 20;11(10):e0162563. doi: 10.1371/journal.pone.0162563. eCollection 2016. PMID 27764102
- [Background] Cairns M, Roca-Feltrer A, Garske T, Wilson AL, Diallo D, Milligan PJ, Ghani AC, Greenwood BM. Estimating the potential public health impact of seasonal malaria chemoprevention in African children. Nat Commun. 2012 Jun 6;3:881. doi: 10.1038/ncomms1879. PMID 22673908
- [Background] Penny MA, Verity R, Bever CA, Sauboin C, Galactionova K, Flasche S, White MT, Wenger EA, Van de Velde N, Pemberton-Ross P, Griffin JT, Smith TA, Eckhoff PA, Muhib F, Jit M, Ghani AC. Public health impact and cost-effectiveness of the RTS,S/AS01 malaria vaccine: a systematic comparison of predictions from four mathematical models. Lancet. 2016 Jan 23;387(10016):367-375. doi: 10.1016/S0140-6736(15)00725-4. Epub 2015 Nov 6. PMID 26549466
- [Background] Neafsey DE, Juraska M, Bedford T, Benkeser D, Valim C, Griggs A, Lievens M, Abdulla S, Adjei S, Agbenyega T, Agnandji ST, Aide P, Anderson S, Ansong D, Aponte JJ, Asante KP, Bejon P, Birkett AJ, Bruls M, Connolly KM, D'Alessandro U, Dobano C, Gesase S, Greenwood B, Grimsby J, Tinto H, Hamel MJ, Hoffman I, Kamthunzi P, Kariuki S, Kremsner PG, Leach A, Lell B, Lennon NJ, Lusingu J, Marsh K, Martinson F, Molel JT, Moss EL, Njuguna P, Ockenhouse CF, Ogutu BR, Otieno W, Otieno L, Otieno K, Owusu-Agyei S, Park DJ, Pelle K, Robbins D, Russ C, Ryan EM, Sacarlal J, Sogoloff B, Sorgho H, Tanner M, Theander T, Valea I, Volkman SK, Yu Q, Lapierre D, Birren BW, Gilbert PB, Wirth DF. Genetic Diversity and Protective Efficacy of the RTS,S/AS01 Malaria Vaccine. N Engl J Med. 2015 Nov 19;373(21):2025-2037. doi: 10.1056/NEJMoa1505819. Epub 2015 Oct 21. PMID 26488565
- [Background] Swysen C, Vekemans J, Bruls M, Oyakhirome S, Drakeley C, Kremsner P, Greenwood B, Ofori-Anyinam O, Okech B, Villafana T, Carter T, Savarese B, Duse A, Reijman A, Ingram C, Frean J, Ogutu B; Clinical Trials Partnership Committee. Development of standardized laboratory methods and quality processes for a phase III study of the RTS, S/AS01 candidate malaria vaccine. Malar J. 2011 Aug 4;10:223. doi: 10.1186/1475-2875-10-223. PMID 21816032
- [Background] Plowe CV, Djimde A, Bouare M, Doumbo O, Wellems TE. Pyrimethamine and proguanil resistance-conferring mutations in Plasmodium falciparum dihydrofolate reductase: polymerase chain reaction methods for surveillance in Africa. Am J Trop Med Hyg. 1995 Jun;52(6):565-8. doi: 10.4269/ajtmh.1995.52.565. PMID 7611566
- [Background] Djimde A, Doumbo OK, Cortese JF, Kayentao K, Doumbo S, Diourte Y, Coulibaly D, Dicko A, Su XZ, Nomura T, Fidock DA, Wellems TE, Plowe CV. A molecular marker for chloroquine-resistant falciparum malaria. N Engl J Med. 2001 Jan 25;344(4):257-63. doi: 10.1056/NEJM200101253440403. PMID 11172152
- [Background] Djimde AA, Fofana B, Sagara I, Sidibe B, Toure S, Dembele D, Dama S, Ouologuem D, Dicko A, Doumbo OK. Efficacy, safety, and selection of molecular markers of drug resistance by two ACTs in Mali. Am J Trop Med Hyg. 2008 Mar;78(3):455-61. PMID 18337343
- [Background] Cairns M, Cheung YB, Xu Y, Asante KP, Owusu-Agyei S, Diallo D, Konate AT, Dicko A, Chandramohan D, Greenwood B, Milligan P. Analysis of Preventive Interventions for Malaria: Exploring Partial and Complete Protection and Total and Primary Intervention Effects. Am J Epidemiol. 2015 Jun 15;181(12):1008-17. doi: 10.1093/aje/kwv010. Epub 2015 May 27. PMID 26022663
- [Background] Xu Y, Cheung YB, Lam KF, Milligan P. Estimation of summary protective efficacy using a frailty mixture model for recurrent event time data. Stat Med. 2012 Dec 20;31(29):4023-39. doi: 10.1002/sim.5458. Epub 2012 Jul 5. PMID 22764039
- [Result] Chandramohan D, Zongo I, Sagara I, Cairns M, Yerbanga RS, Diarra M, Nikiema F, Tapily A, Sompougdou F, Issiaka D, Zoungrana C, Sanogo K, Haro A, Kaya M, Sienou AA, Traore S, Mahamar A, Thera I, Diarra K, Dolo A, Kuepfer I, Snell P, Milligan P, Ockenhouse C, Ofori-Anyinam O, Tinto H, Djimde A, Ouedraogo JB, Dicko A, Greenwood B. Seasonal Malaria Vaccination with or without Seasonal Malaria Chemoprevention. N Engl J Med. 2021 Sep 9;385(11):1005-1017. doi: 10.1056/NEJMoa2026330. Epub 2021 Aug 25. PMID 34432975
- [Derived] Ali MS, Stockdale L, Sagara I, Zongo I, Yerbanga RS, Mahamar A, Nikiema F, Tapily A, Sompougdou F, Diarra M, Bellamy D, Provstgaard-Morys S, Zoungrana C, Issiaka D, Haro A, Sanogo K, Sienou AA, Kaya M, Traore S, Dicko OM, Kone Y, Yalcouye H, Thera I, Diarra K, Snell P, Ofori-Anyinam O, Ockenhouse C, Lee C, Ewer K, Tinto H, Djimde A, Ouedraogo JB, Dicko A, Chandramohan D, Greenwood B. The anti-circumsporozoite antibody response to repeated, seasonal booster doses of the malaria vaccine RTS,S/AS01E. NPJ Vaccines. 2025 Feb 6;10(1):26. doi: 10.1038/s41541-025-01078-0. PMID 39915506
- [Derived] Cairns M, Barry A, Zongo I, Sagara I, Yerbanga SR, Diarra M, Zoungrana C, Issiaka D, Sienou AA, Tapily A, Sanogo K, Kaya M, Traore S, Diarra K, Yalcouye H, Sidibe Y, Haro A, Thera I, Snell P, Grant J, Tinto H, Milligan P, Chandramohan D, Greenwood B, Dicko A, Ouedraogo JB. The duration of protection against clinical malaria provided by the combination of seasonal RTS,S/AS01E vaccination and seasonal malaria chemoprevention versus either intervention given alone. BMC Med. 2022 Oct 7;20(1):352. doi: 10.1186/s12916-022-02536-5. PMID 36203149
- [Derived] Grant J, Sagara I, Zongo I, Cairns M, Yerbanga RS, Diarra M, Zoungrana C, Issiaka D, Nikiema F, Sompougdou F, Tapily A, Kaya M, Haro A, Sanogo K, Sienou AA, Traore S, Thera I, Yalcouye H, Kuepfer I, Snell P, Milligan P, Ockenhouse C, Ofori-Anyinam O, Tinto H, Djimde A, Chandramohan D, Greenwood B, Dicko A, Ouedraogo JB. Impact of seasonal RTS,S/AS01E vaccination plus seasonal malaria chemoprevention on the nutritional status of children in Burkina Faso and Mali. Malar J. 2022 Feb 22;21(1):59. doi: 10.1186/s12936-022-04077-x. PMID 35193608
- [Derived] Sagara I, Zongo I, Cairns M, Yerbanga RS, Mahamar A, Nikiema F, Tapily A, Sompougdou F, Diarra M, Zoungrana C, Issiaka D, Haro A, Sanogo K, Aziz Sienou A, Kaya M, Traore S, Thera I, Diarra K, Dolo A, Kuepfer I, Snell P, Milligan P, Ockenhouse C, Ofori-Anyinam O, Tinto H, Djimde A, Ouedraogo JB, Dicko A, Chandramohan D, Greenwood B. The Anti-Circumsporozoite Antibody Response of Children to Seasonal Vaccination With the RTS,S/AS01E Malaria Vaccine. Clin Infect Dis. 2022 Sep 10;75(4):613-622. doi: 10.1093/cid/ciab1017. PMID 34894221
- [Derived] Chandramohan D, Dicko A, Zongo I, Sagara I, Cairns M, Kuepfer I, Diarra M, Tapily A, Issiaka D, Sanogo K, Mahamar A, Sompougdou F, Yerbanga S, Thera I, Milligan P, Tinto H, Ofori-Anyinam O, Ouedraogo JB, Greenwood B. Seasonal malaria vaccination: protocol of a phase 3 trial of seasonal vaccination with the RTS,S/AS01E vaccine, seasonal malaria chemoprevention and the combination of vaccination and chemoprevention. BMJ Open. 2020 Sep 15;10(9):e035433. doi: 10.1136/bmjopen-2019-035433. PMID 32933955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 PLUS SMC With SP+AQ
Started | 1965 | 1988 | 1967
Completed | 1716 | 1734 | 1740
Not Completed | 249 | 254 | 227

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 PLUS SMC With SP+AQ | Total
Number analyzed (Participants) | 1965 | 1988 | 1967 | 5920
Age, Customized [Count of Participants; unit: Participants] — Age at first vaccination
  Participants
    Under 8 months | 471 | 448 | 463 | 1382
    8-11 months | 532 | 527 | 531 | 1590
    12-15 months | 486 | 552 | 537 | 1575
    16 months or older | 476 | 461 | 436 | 1373
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 950 | 956 | 948 | 2854
  Male | 1015 | 1032 | 1019 | 3066
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 936 | 911 | 930 | 2777
  Mali | 1029 | 1077 | 1037 | 3143
LLIN use the night before the 2017 census [Count of Participants; unit: Participants] — LLIN - Long-lasting Insecticide Treated Net
  Participants
    Yes | 1593 | 1580 | 1577 | 4750
    No | 360 | 391 | 380 | 1131
    Missing | 12 | 17 | 10 | 39
PCV vaccination [Count of Participants; unit: Participants] — PCV- 11 valent pneumococcal conjugate vaccine
  Participants
    Yes | 1650 | 1646 | 1642 | 4938
    No | 82 | 99 | 74 | 255
    Card not available | 172 | 175 | 171 | 518
    Card available but incomplete | 61 | 67 | 79 | 207
    Missing | 0 | 1 | 1 | 2
Penta vaccination [Count of Participants; unit: Participants] — Penta vaccine - tetanus, diphtheria, hepatitis B and Hemophilus influenzae type b conjugate vaccine
  Participants
    Yes | 1650 | 1647 | 1650 | 4947
    No | 87 | 95 | 78 | 260
    Card not available | 169 | 179 | 167 | 515
    Card available but incomplete | 58 | 66 | 67 | 191
    Missing | 1 | 1 | 5 | 7
MenAfriVac vaccination [Count of Participants; unit: Participants] — MenAfriVac - group A meningococcal conjugate vaccine
  Participants
    Yes | 468 | 477 | 478 | 1423
    No | 1245 | 1251 | 1251 | 3747
    Missing | 252 | 260 | 238 | 750

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Episodes of Malaria
Description: Passive surveillance to detect episode of fever (temperature > 37.5 C), or a history of fever within the past 48 hours, that is severe enough to require treatment at a health centre and which is accompanied by a positive blood film with a parasite density of 5,000 per µl or more
Time Frame: Passive surveillance of clinical episodes of malaria within the study area starting from the date of the first dose of study vaccines (April/May 2017) until 31st March 2020- a total of 36 months.
Measure: Number (95% Confidence Interval); unit: No. of events/1000 person years at risk
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 PLUS SMC With SP+AQ
Number analyzed (Participants) | 1965 | 1988 | 1967
No. of events/1000 person years at risk | 304.8 [290.5 to 319.8] | 278.2 [264.6 to 292.4] | 113.3 [104.7 to 122.5]

2. Secondary Outcome: Clinical Episodes of Uncomplicated Febrile Illness
Description: Passive and active surveillance to detect cases with temperature > 37.5o C), or a history of fever within the past 48 hours, with a positive blood film (any level of asexual parasitaemia) or a positive rapid diagnostic test (RDT) for malaria
Time Frame: Passive surveillance in all health centers within the study area, active surveillance in a sub set of study children starting July 2017 till April 2020.
Reporting Status: Not Posted

3. Secondary Outcome: Hospital Admissions With Malaria, Including Severe Malaria
Description: Hospital admissions with malaria, including cases of severe malaria which meet WHO criteria for a diagnosis of severe malaria.
Time Frame: Through study completion (30 months), each child admitted in a study hospital will be treated and monitored until complete cure or death (a period of 3 years). Documentation of each hospital admission according to ICH-GCP.
Reporting Status: Not Posted

4. Secondary Outcome: Prevalence of Malaria Infection Not Severe Enough to Warrant a Clinic Visit
Description: Active surveillance of malaria at household level to assess the prevalence of malaria infection not severe enough to warrant a clinic visit detected in a subset of randomly selected children.
Time Frame: Weekly home visits through study completion from July 2017 - April 2020 to screen study children for malaria.
Reporting Status: Not Posted

5. Secondary Outcome: Prevalence of Malaria Parasitaemia, Including Gametocytaemia and the Prevalence of Moderate and Severe Anemia and Malnutrition
Description: The prevalence of malaria parasitaemia, including gametocytaemia, moderate and severe anaemia and malnutrition at the end of the malaria transmission season
Time Frame: Blood sample collection during 2-week cross sectional survey at the end of each malaria transmission season.
Reporting Status: Not Posted

6. Secondary Outcome: Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs), including any deaths, occurring at any time during the study with special reference to any cases of meningitis and cerebral malaria (WHO case definition)
Time Frame: Through study completion (for 30 months), each SAE will be treated and documented according to ICH-GCP.
Reporting Status: Not Posted

7. Secondary Outcome: Immune Response to the Vaccine (Anti-CSP Antibody Concentrations)
Description: After priming and after each booster dose, determined in a sub-sample of children
Time Frame: Blood sample collection prior to 1st dose of vaccine and 1 month after 3rd dose of the primary series of vaccination. In years 2 and 3 blood will be collected before the booster dose and 1 month after administration of the 4th (and 5th) vaccine dose.
Reporting Status: Not Posted

8. Secondary Outcome: Drug Resistance to SP and AQ
Description: The presence of molecular markers of resistance to SP and AQ in parasite positive samples
Time Frame: Blood sample collection during the 2-week cross sectional survey conducted at the end of malaria transmission season in 2019.
Reporting Status: Not Posted

9. Secondary Outcome: Prevalence of Malaria Parasitaemia in School Aged Children
Description: The prevalence of malaria parasitaemia at the end of the malaria transmission season in school-age children resident in the study areas, to determine overall malaria transmission
Time Frame: Blood sample collection during the 2-week cross sectional survey at the end of the malaria transmission season in Year 2 and 3 (November 2018/19).
Reporting Status: Not Posted

10. Secondary Outcome: SP+AQ Drug Sensitivity
Description: The 28-day treatment outcome in children with asymptomatic malaria parasitaemia treated with SP+AQ.
Time Frame: Children with asymptomatic malaria parasitaemia identified during the final cross-sectional survey (November 2019), treated with a full course of SP+AQ over 3 days and followed for 28 days.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Acceptability of RTS,S and SMC
Description: The acceptability of the two interventions (separately and combined) to the health care deliverers and to the study communities (standardized questionnaires)
Time Frame: Data collection in Year 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Feasibility of Introducing Two Malaria Control Strategies Simultaneously
Description: The feasibility of introducing two malaria control strategies simultaneously from the health system perspective (structured observations and interviews with health system officials)
Time Frame: Data collection in Year 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious adverse event data were collected over a 3 year period, from 1st April 2017 to 31st March 2020.
Description: The number of participants at risk for other (non-serious) adverse events is zero because non-serious adverse events were not collected or assessed as part of this study.
Arm/Group | SMC With SP+AQ | RTS,S/AS01 | RTS,S/AS01 PLUS SMC With SP+AQ
All-Cause Mortality (participants affected / at risk) | 32/1965 | 27/1988 | 15/1967
Serious Adverse Events (participants affected / at risk) | 97/1965 | 94/1988 | 71/1967
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMC With SP+AQ (N=1965) | RTS,S/AS01 (N=1988) | RTS,S/AS01 PLUS SMC With SP+AQ (N=1967)
Non-fatal SAEs (General disorders) | 65 | 67 | 56
Fatal SAEs (General disorders) | 32 | 27 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03143218/Prot_SAP_000.pdf